CLINICAL TRIAL: NCT01669889
Title: A Multi-center, Non-drug Study to Explore the Relationship Between Exploratory Biomarkers and Functional Dimensions in Individuals With Autistic Disorder or Asperger's Syndrome.
Brief Title: A Non-Drug Study on the Relationship Between Exploratory Biomarkers and Functional Dimensions in Individuals With Autistic Disorder or Asperger's Syndrome
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BP28421
Record Dates: First submitted 2012-08-15; First posted 2012-08-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer, Autistic Disorder, Asperger's Syndrome
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center, non-drug study will explore the relationship between exploratory biomarkers and functional dimensions in male adult individuals with Autistic Disorder or Asperger's Syndrome and healthy volunteer controls. Subjects will undergo a number of assessments on study visit Day 1.

ELIGIBILITY:
Inclusion Criteria:

Individuals with Autistic Disorder or Asperger's Syndrome:

* Male adults, 18 to 45 years of age inclusive
* Diagnosis of Autistic Disorder or Asperger's Syndrome as defined by DSM-IV
* IQ >70
* Body mass index (BMI) 18 to 35 kg/m2
* Availability of a reliable caregiver, able and willing to provide information regarding the individual's behavior and symptoms

Healthy controls:

* Healthy male adults, 18 to 45 years of age inclusive
* IQ >70
* Body mass index (BMI) 18 to 30 kg/m2

Exclusion Criteria:

General exclusion criteria:

* Positive test for drugs of abuse or alcohol
* Confirmed systolic blood pressure >140 or <90 mmHg, and diastolic blood pressure >90 or <50 mmHg
* Resting pulse rate >100 or <40 beats per minute
* Alcohol and/or substance abuse/dependence during the last 12 months
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study

Additionally for individuals with Autistic Disorder or Asperger's Syndrome:

* History of epilepsy/seizure disorder (except simple febrile seizures)

  * Significant disruptive, aggressive or self-injurious, or sexually inappropriate behavior during the last 3 months that in the opinion of the investigator might interfere with the conduct of the study

Additionally for healthy controls:

* Clinically significant abnormalities in laboratory test results
* History of or current psychiatric, neurological disorder or pervasive developmental disorder

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: High functioning (IQ >70) male adult individuals with Autistic Disorder or Asperger's Syndrome and age and IQ matched healthy male volunteers
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Behavior assessment ratings | approximately 5 months
Cognition assessment ratings | approximately 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - Los Ageles, California
  - New Haven, Connecticut
  - New York, New York